CLINICAL TRIAL: NCT02607176
Title: A Post -Marketing Drug Evaluation(Phase IV Clinical Trial) to Study the Safety and Efficacy of Heweizhixie Capsule in Patients With Diarrhea
Brief Title: Heweizhixie capsuleTherapy on Patients With Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Longhua Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZY3-CCCX-3-1001
Record Dates: First submitted 2015-11-14; First posted 2015-11-17 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heweizhixie capsule (Experimental): Heweizhixie capsule, 0.33g/#, 3 #, Tid, Oral
  Interventions: Drug: Heweizhixie capsule

INTERVENTIONS:
Drug: Heweizhixie capsule — 3 #, Tid, Oral for 3 days
  Other Names: Changdaoqing capsule

SUMMARY:
The objective of this study is to evaluate safety and efficacy of Heweizhixie Capsule in patients with diarrhea.

DETAILED DESCRIPTION:
The objective of this study is to evaluate safety and efficacy of Heweizhixie Capsule in patients with diarrhea.This is a Phase 4 Open Label trial, enroll 2400 patients with diarrhea Primary Outcome Measure:Percent of subjects with treatment Success

Secondary Outcome Measures:

Number of unformed stools passed per 24 h period Time (hours) from first intake to the last unformed stools Change from baseline of Leeds dyspepsia questionnaire score Percent of subjects with AE.

ELIGIBILITY:
Inclusion Criteria:

3 or more unformed stools in 24 hours Male and female subjects between 18 and 80 years old Signed informed consent

Exclusion Criteria:

Subjects with serum ALT more than 5ULN or serum Cr more than 442umol/L Subjects are pregnant now, likely to become pregnant Subjects, who in the opinion of the Investigator, are not suitable candidates for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with treatment Success | 3 days
  Percent of subjects with treatment Success

SECONDARY OUTCOMES:
Number of unformed stools passed per 24 h period | per 24 h period
  Number of unformed stools passed per 24 h period
Time (hours) from first intake to the last unformed stools | 3 days
  Time (hours) from first intake to the last unformed stools
Change from baseline of leeds dyspepsia questionnaire score | 3 days
  Change from baseline of leeds dyspepsia questionnaire score
Percent of subjects with AE | 3 days
  Percent of subjects with AE

CONTACTS AND LOCATIONS:
Overall Officials: QingShan Zheng, Dr, Study Chair — Shanghai University of Chinese Medicine
Locations (1):
- Long hua hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No